CLINICAL TRIAL: NCT07119983
Title: Effect of Stress Ball Applied During Surgical Debridement/Dressing on Pain, Distress, and Physiological Parameters in Patients With Diabetic Foot Ulcers: A Randomized Controlled Trial
Brief Title: Effect of Stress Ball Applied During Surgical Debridement/Dressing on Pain, Distress, and Physiological Parameters in Patients With Diabetic Foot Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Derya Gezer, Assistant Professor, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Stress Ball
Record Dates: First submitted 2025-07-28; First posted 2025-08-13 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot Ulcer Associated With Type II Diabetes Mellitus
Keywords: Diabetic foot ulcer; sharp debridement; pain; anxiety; stress ball; nursing care
MeSH Terms: conditions — Diabetic Foot; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled experimental design aimed at evaluating the effects of stress ball use on pain, anxiety, distress, and physiological parameters during surgical debridement in individuals with diabetic foot ulcers.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress ball (Experimental): The effects of stress balls on pain, distress and physiological parameters during surgical debridement in patients with diabetic foot ulcers will be investigated.
  Interventions: Behavioral: Stress ball
- Control Group (No Intervention): Routine care

INTERVENTIONS:
Behavioral: Stress ball — The effects of stress balls on pain, distress and physiological parameters during surgical debridement in patients with diabetic foot ulcers will be investigated.
  Arms: Stress ball

SUMMARY:
Diabetes mellitus (DM) is a common metabolic disease characterized by hyperglycemia, resulting from a deficiency or insufficiency of insulin. Diabetic foot ulcers (DFU), a late complication of diabetes, develop as a result of peripheral neuropathy, peripheral arterial disease, and trauma, negatively impacting individuals' quality of life and increasing the rate of hospitalization and amputation. While sharp debridement, one of the most effective methods in the management of diabetic foot ulcers, accelerates healing, it often causes pain and anxiety, which negatively impacts the treatment process. The physiological effects of anxiety include increased respiratory and heart rates, increased blood pressure, and prolonged procedure times. These effects can reduce patient compliance and complicate nursing care.

Non-pharmacological interventions offer important alternatives for pain and anxiety management. One such method, the use of a stress ball, is based on a distraction technique and is used to reduce individuals' emotional and physiological stress levels. The literature has demonstrated the positive effects of stress balls during endoscopy, biopsy, and skin procedures. However, there is insufficient evidence regarding the use of stress balls during sharp debridement. Therefore, this study aimed to evaluate the effects of stress balls on pain, distress, and physiological parameters during surgical debridement in patients with diabetic foot ulcers. The results of this study are expected to contribute to nursing care.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in the study and sign the Informed Consent
* Form will be included in the study.
* They are over 18 years of age,
* They are literate in Turkish,
* They are undergoing surgical debridement for the first time,
* They are receiving inpatient treatment in the ward, and
* They have pain ≥1 on the Visual Analog Scale (VAS) before the procedure.

Exclusion Criteria:

* Patients who have a diagnosed psychiatric or mental illness,
* Regular painkiller use and chronic pain,
* Visual, hearing, perception, or communication problems,
* Physically impaired (such as an open wound on the hand or lack of muscle strength to squeeze a stress ball),
* Decided to undergo an intervention to reduce pain before debridement (such as local anesthesia, nerve blockade, opioid analgesics, etc.),
* Used non-pharmacological methods to reduce pain before the procedure will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | Before the Procedure, during the Procedure (10th minute), and baseline, after an average of 20-30 minutes
  Visual Analogue Scale -VAS: The scale was developed by Price and colleagues in 1983 for use in assessing subjectively perceived pain. Eti-Aslan noted in his study that the VAS is more sensitive and better defined in assessing acute pain. It is a 10 cm (100 mm) ruler with the word "painlessness" written on one end and "the most severe pain" written on the other. Participants were asked to indicate the intensity of pain they were currently experiencing, explaining that "0" on the scale means "I feel no pain" and that increasing numbers indicate increased pain intensity. "10" means "I feel the most severe pain." A higher score on the scale indicates increased pain.
Anxiety Assesment (The Distress Thermometer) | Before the Procedure and baseline, after an average of 20-30 minutes
  The Distress Thermometer was first developed by Roth and colleagues for use in identifying non-pathological distress in patients undergoing cancer treatment after answering the necessary questions. The distress level is rated from 0 to 10. The practitioner expresses the distress experienced using the numbers on the thermometer. A score of zero indicates no distress, while a score of 10 indicates the highest level of distress. The green zone encompasses scores from 0 to 3. Individuals experiencing distress within this range are capable of managing their distress. The yellow zone encompasses scores from 4 to 6. A distress score in this range indicates that the individual is unable to manage their distress and requires intervention to return them to the green zone. The red zone encompasses scores from 7 to 10. Individuals experiencing distress within this range require urgent and comprehensive intervention.
Physiological Parameters (heart rate, systolic and diastolic blood pressure, oxygen saturation and respiratory rate) | Before the Procedure, during the Procedure (10th minute), and baseline, after an average of 20-30 minutes
  Heart rate, systolic and diastolic blood pressure, oxygen saturation, and respiratory rate will be recorded before, during, and after debridement. Systolic and diastolic blood pressure will be measured for patients in the study and control groups using the ERKA adult aneroid blood pressure monitor, while oxygen saturation and heart rate will be measured using the Masimo SET® Pulse Oximetry. Both devices will be calibrated before data collection.
Physiological Parameter: heart rate | Before the Procedure, during the Procedure (10th minute), and baseline, after an average of 20-30 minutes
  Heart rate will be measured using the Masimo SET® Pulse Oximetry. Devices will be calibrated before data collection.
Physiological Parameters: systolic and diastolic blood pressure | Before the Procedure, during the Procedure (10th minute), and baseline, after an average of 20-30 minutes
  Systolic and diastolic blood pressure will be measured for patients in the study and control groups using the ERKA adult aneroid blood pressure monitor
Physiological Parameter: oxygen saturation | Before the Procedure, during the Procedure (10th minute), and baseline, after an average of 20-30 minutes
  Oxygen saturation will be measured using the Masimo SET® Pulse Oximetry. Device will be calibrated before data collection.
Physiological Parameter: respiratory rate | Before the Procedure, during the Procedure (10th minute), and baseline, after an average of 20-30 minutes
  Respiratory rate will be monitored for one minute, with each inspiration and expiration counted as a breath.

OTHER OUTCOMES:
Meggitt-Wagner classification | in recruitment
  Meggitt-Wagner Classification of Diabetic Foot:
  The Meggitt-Wagner classification was developed by Meggitt in 1976 and revised by Wagner in 1981. This classification system, which grades the wound into six categories from stage 0 to stage 5 based on the depth of the wound and the presence of osteomyelitis and gangrene, is evaluated based on observational findings, excluding ulcer depth. Findings of ischemia and infection are limited and do not include the presence of neuropathy. However, evaluation of these factors is known to have a positive impact on the healing process of diabetic foot ulcers.

CONTACTS AND LOCATIONS:
Overall Officials: DERYA GEZER, Asisstant Professor, Study Chair — Tarsus University; EZGİ MUTLUAY YAYLA, Asisstant Professor, Study Director — Tarsus University; DUDU ALPTEKİN, Dr, Study Director — CUKUROVA UNİVERSİTY
Locations (1):
- Tarsus University, Mersin, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Results regarding the effects of stress ball use on pain, anxiety, and hemodynamic parameters surgical debridement in individuals with diabetic foot ulcers will be shared. However, your personal information will not be shared.
Supporting Information: CSR

REFERENCES:
- [Background] Purcell A, Buckley T, King J, Moyle W, Marshall AP. Topical Analgesic and Local Anesthetic Agents for Pain Associated with Chronic Leg Ulcers: A Systematic Review. Adv Skin Wound Care. 2020 May;33(5):240-251. doi: 10.1097/01.ASW.0000658572.14692.fb. PMID 32304447
- [Background] Hajimohammadi K, Parizad N, Bagheri M, Faraji N, Goli R. Maggot therapy, alginate dressing, and surgical sharp debridement: Unique path to save unresponsive diabetic foot ulcer. Int J Surg Case Rep. 2023 Oct;111:108907. doi: 10.1016/j.ijscr.2023.108907. Epub 2023 Oct 4. PMID 37804682
- [Background] Shamloul G, Khachemoune A. Reappraisal and updated review of maggot debridement therapy in chronic lower extremity ulcers. Int J Dermatol. 2023 Jul;62(7):962-968. doi: 10.1111/ijd.16619. Epub 2023 Mar 7. PMID 36880424
- [Background] McDermott K, Fang M, Boulton AJM, Selvin E, Hicks CW. Etiology, Epidemiology, and Disparities in the Burden of Diabetic Foot Ulcers. Diabetes Care. 2023 Jan 1;46(1):209-221. doi: 10.2337/dci22-0043. PMID 36548709
- [Background] Sriubolmas N, Panbangred W, Sriurairatana S, Meevootisom V. Localization and characterization of inclusion bodies in recombinant Escherichia coli cells overproducing penicillin G acylase. Appl Microbiol Biotechnol. 1997 Apr;47(4):373-8. doi: 10.1007/s002530050943. PMID 9163951
- [Background] Alshammari L, O'Halloran P, McSorley O, Doherty J, Noble H. The effectiveness of foot care educational interventions for people living with diabetes mellitus: An umbrella review. J Tissue Viability. 2023 Aug;32(3):406-416. doi: 10.1016/j.jtv.2023.06.001. Epub 2023 Jun 16. PMID 37369610
- [Background] van Netten JJ, Raspovic A, Lavery LA, Monteiro-Soares M, Paton J, Rasmussen A, Sacco ICN, Bus SA. Prevention of foot ulcers in persons with diabetes at risk of ulceration: A systematic review and meta-analysis. Diabetes Metab Res Rev. 2024 Mar;40(3):e3652. doi: 10.1002/dmrr.3652. Epub 2023 May 27. PMID 37243880
- [Background] Aslan F, Tosun B, Altinok Ersoy N, Ozen N. The effect of a stress ball on pain and anxiety during sharp debridement in patients with diabetic foot ulcers: A randomized controlled, single-blind study. J Tissue Viability. 2025 May;34(2):100861. doi: 10.1016/j.jtv.2025.100861. Epub 2025 Jan 26. PMID 39892227
- [Background] Najafi B, Mishra R. Harnessing Digital Health Technologies to Remotely Manage Diabetic Foot Syndrome: A Narrative Review. Medicina (Kaunas). 2021 Apr 14;57(4):377. doi: 10.3390/medicina57040377. PMID 33919683
- [Background] Yang L, Rong GC, Wu QN. Diabetic foot ulcer: Challenges and future. World J Diabetes. 2022 Dec 15;13(12):1014-1034. doi: 10.4239/wjd.v13.i12.1014. PMID 36578870